CLINICAL TRIAL: NCT03200756
Title: The Effect of Cardiac Rehabilitation on Sedentary Behavior
Brief Title: Cardiac Rehabilitation and Sedentary Behavior
Acronym: Rest-CR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-1914
Record Dates: First submitted 2017-06-21; First posted 2017-06-27 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Cardiovascular Diseases
Keywords: sedentary behavior
MeSH Terms: conditions — Cardiovascular Diseases; Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sedentary Group (Experimental): The experimental group undergoes a behavioral intervention to reduce sedentary behavior which includes a patient centered approach with monitoring and goal setting.
  Interventions: Behavioral: Sedentary Group
- Exercise Group (Active Comparator): The Active Comparative group undergoes a standard clinical approach to increase exercise which is patient centered with monitoring and goal setting.
  Interventions: Behavioral: Exercise Group

INTERVENTIONS:
Behavioral: Sedentary Group — The sedentary group undergoes a behavioral intervention to reduce sedentary behavior which includes a patient centered approach with monitoring and goal setting.
  Arms: Sedentary Group
Behavioral: Exercise Group — The Active Comparative group undergoes a standard clinical approach to increase exercise which is patient centered with monitoring and goal setting.
  Arms: Exercise Group

SUMMARY:
This trial randomizes patients who plan to attend cardiac rehabilitation to either a behavioral intervention to specifically reduce sedentary behavior or to usual care which exclusively focuses on increasing exercise.

DETAILED DESCRIPTION:
Cardiac rehabilitation after a cardiac event or procedure is of key importance to physical and psychological recovery. Cardiac rehabilitation comprises a standardized stepwise approach to exercise in a supervised setting and is proven to reduce morbidity and mortality after a cardiac event. However, cardiac rehabilitation does not necessarily change behavior in the long-term and many do not attend cardiac rehabilitation due to lack of motivation, difficulty accessing programs, and cost. These individuals loose an important opportunity to improve their health, sense of well-being and outcomes. The investigators propose to test the effect of a patient-centered approach to reduce sedentary behavior for aging adults added to usual cardiac rehabilitation. In this study, the investigators will identify patients at their introductory visit to cardiac rehabilitation and randomize to either a program to decrease in-home sedentary behavior vs. a standard program to increase in-home exercise. Both groups will receive additional support and encouragement to attend cardiac rehabilitation. Using motivational interviewing techniques in both groups the investigators will assist the patients in recognizing their potential and goal-setting. Patients will be monitored using the ActivPAL monitor, a new technology that quantifies sedentary time and steps/day. Patients will be monitored four times as they proceed through cardiac rehabilitation for a total of 13 weeks and receive 3 educational and goal setting sessions. Those in the intervention group will have sedentary behavior change emphasized with feedback from the ActivPAL monitor. The control group will focus on standard exercise recommendations and feedback from his/her exercise diary. Outcomes include change in sedentary time and steps/day. Anticipated results include a significant change in the intervention group vs. the control: a decrease in in-home sedentary time, an increase in steps/day. The results of this study will provide the basis for designing a larger randomized controlled trial to investigate the effects of an intervention to reduce sedentary behavior as an adjunct to cardiac rehabilitation especially for older adults. Additional investigation will be warranted for those who do not attend cardiac rehabilitation but are able to follow a post-cardiac event program to reduce in-home sedentary behavior.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in Cardiac Rehabilitation
* Age 50 years old or greater
* Short Physical Performance Battery (SPPB) score equal or less than 10

Exclusion Criteria:

* Hypoxia
* Orthopedic Disease that limits mobility
* Neurologic Disease that limits mobility
* Metastatic Cancer
* Life expectancy of <6 months
* Depression
* Montreal Cognitive Assessment less than 24
* Left Ventricular Assist Device (LVAD)
* Cardiac Transplant
* Patient Health Questionnaire-9 (PHQ-9) of 15 or greater

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2017-06-20 (Actual)

PRIMARY OUTCOMES:
Change in steps per day from before to after cardiac rehabilitation | 1 full week of Activpal data collected at week1, week 7, week 13, week 17 of the study
  The number of steps per day will be recorded using the Activpal monitor. Investigators will compare the number of steps per day prior to the subject beginning rehabiliation to the number of steps per day after cardiac rehabilitation is complete
Change in sedentary time from before to after cardiac rehabilitation | 1 full week of Activpal data collected at week1, week 7, week 13, week 17 of the study
  The number of sedentary hours per day will be recorded using the Activpal monitor.Investigators will compare the number of sedentary hours per day recorded prior to the subject beginning cardiac rehabilitation to the number of sedentary hours per day recorded after cardiac rehabilitation is complete

CONTACTS AND LOCATIONS:
Overall Officials: Boxer Rebecca, MD,MS, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital Cardiovascular Rehabilitation, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No